CLINICAL TRIAL: NCT04461210
Title: Objective Assessment of Pain Thresholds in Women With Vulvodynia
Brief Title: Vulvodynia Pain Thresholds
Status: Terminated | Type: Observational
Why Stopped: Investigator retired and no other investigator was able to resume the study.
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Vanessa Barnabei, Professor, State University of New York at Buffalo
Other Study IDs: 00004558; UL1TR001412 (NIH)
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vulvodynia: Women with localized, provoked vulvodynia
  Interventions: Diagnostic Test: Thermographic Imaging and Mechanical Pain Assessment
- Health Controls: Women without vulvar pain or other vulvar disorders.
  Interventions: Diagnostic Test: Thermographic Imaging and Mechanical Pain Assessment

INTERVENTIONS:
Diagnostic Test: Thermographic Imaging and Mechanical Pain Assessment — Assessment of pain sensitivity with mechanical stimulus (cotton swab) and thermographic imaging with infrared camera

SUMMARY:
Annotated pain maps will be created showing region and size of areas sensitive to mechanical stimulus in both women affected by vulvar pain and unaffected control patients.

DETAILED DESCRIPTION:
The investigators will develop annotated pain maps showing region and size of areas sensitive to mechanical stimulus. The pain maps will be created by combining IR images, photographs, and clinical input, and will be correlated with patient co-morbidities. The IR images will assess for areas of inflammation and increased skin temperature. Pain maps will be created with patient response to mechanical stimulation with a cotton swab and will be overlaid on the thermographic images. Through this combination of measurements, the investigators plan to expand the diagnostic tools used in patient care as well as on the classification of this heterogeneous disorder.

ELIGIBILITY:
Inclusion Criteria:

* women meeting criteria for vulvodynia women seeking care for routine gynecologic exam

Exclusion Criteria:

* women less than 18 years of age current pregnancy women with vulvar or vaginal disorder other than pain

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Vulvodynia is a sex-specific disorder. Only women will be enrolled.
Study Population: Women with localized, provoked vulvodynia and healthy controls without vulvar pain or other vulvar disorders.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa M Barnabei, MD, PhD, Principal Investigator — University at Buffalo
Locations (1):
- UBMD Obstetrics and Gynecology, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: Women without vulvar pain or other vulvar disorders.
  Thermographic Imaging and Mechanical Pain Assessment: Assessment of pain sensitivity with mechanical stimulus (cotton swab) and thermographic imaging with infrared camera
Period: Overall Study
Arm/Group | Vulvodynia | Healthy Controls
Started | 4 | 14
Completed | 4 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vulvodynia | Healthy Controls | Total
Number analyzed (Participants) | 4 | 14 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] — mean age of each group
  years | 32 (10) | 30 (9.3) | 30.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 14 | 18
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — No exclusions based on ethnicity.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 4 | 14 | 18
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 11 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 14 | 18

OUTCOME MEASURES:

1. Primary Outcome: Annotated Pain Mapping
Description: Develop annotated pain maps showing region and size of area sensitive to mechanical stimulus. A cotton swab is used to lightly touch the vulva in 18 different locations and participant's assessment of pain on a scale of 0-10 is recorded.
Time Frame: Duration of study visit, approximately 1 hour
Population: Outcome measure is the average of the pain scores (scale 0-10 with 10 being worst) at 7 points of the inner vulva.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Vulvodynia | Healthy Controls
Number analyzed (Participants) | 4 | 14
score on a scale | 4.7 [0 to 10] | 1.9 [0 to 10]

2. Primary Outcome: Quantitative Pain Description of the Vulva With Touch.
Description: The vulva is lightly touched with a cotton swab at 18 locations of the vulva. Participants rate pain at each location on a scale of 0-10, with 0 being no pain and 10 being worst. Only the pain scores from the 7 points of the inner vulva are presented here, since that is the primary site of pain in women with provoked vulvodynia.
Time Frame: Immediate
Population: number of participants assessed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vulvodynia | Health Controls
Number analyzed (Participants) | 4 | 14
score on a scale | 3.5 (4.7) | 1.1 (1.9)

3. Secondary Outcome: Thermographic Imaging of the Vulva.
Description: Images of the vulva taken (prior to any provocation) with specialized temperature-sensitive camera. These images will then be overlaid on the annotated pain map.
Time Frame: Duration of study visit, approximately 1 hour
Population: Maximum and minimum temperature assessment from images of the outer vulva at 12 touch points; Mean +/- SD.
Measure: Mean (Standard Deviation); unit: temperature in Fahrenheit
Arm/Group | Vulvodynia | Health Controls
Number analyzed (Participants) | 4 | 13
temperature in Fahrenheit
  maximum temperature | 36.4 (0.21) | 36.8 (0.58)
  minimum temperature | 32.2 (1.8) | 31.9 (1.65)

4. Secondary Outcome: Thermographic Imaging of the Vulva
Description: Images of the vulva taken with specialized heat-sensitive camera.
Time Frame: Duration of study visit, about 1 hour
Population: Maximum and minimum temperature assessment from images of the inner vulva; Mean +/- SD.
Measure: Mean (Standard Deviation); unit: temperature in Fahrenheit
Arm/Group | Vulvodynia | Health Controls
Number analyzed (Participants) | 4 | 13
temperature in Fahrenheit
  maximum temperature | 36.9 (0.47) | 37.4 (0.47)
  minimum temperature | 33.2 (1.8) | 34.3 (2.1)

ADVERSE EVENTS:
Time Frame: Event reporting occurred for the duration of the participant's time in the study, generally about 1 hour.
Description: This was an observational study with no intervention and essentially no risk for serious adverse events. Temporary discomfort with touch of the cotton swab during examination, especially in participants with known history of vulvar pain, was expected. No participant noted persistent or worsening pain following the examination.
Groups:
- Vulvodynia: Women with localized, provoked vulvodynia
  Thermographic Imaging and Mechanical Pain Assessment: Assessment of pain sensitivity with mechanical stimulus (cotton swab) and thermographic imaging with infrared camera
  No adverse events.
- Healthy Controls: Women without vulvar pain or other vulvar disorders.
  Thermographic Imaging and Mechanical Pain Assessment: Assessment of pain sensitivity with mechanical stimulus (cotton swab) and thermographic imaging with infrared camera
  No adverse events.
Arm/Group | Vulvodynia | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/14
Other Adverse Events (participants affected / at risk) | 0/4 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT04461210/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT04461210/ICF_001.pdf